CLINICAL TRIAL: NCT01639378
Title: Impact of Renal Artery Denervation in Patients With Chronic Heart Failure Compared With Sham Procedure
Brief Title: Renal Artery Denervation in Chronic Heart Failure Study
Acronym: REACH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REACH
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Systolic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Subjects are treated with renal denervation after randomisation and maintained on heart failure medications
  Interventions: Procedure: Renal Denervation
- Control group (No Intervention): Subject will have a sham procedure and not receive renal denervation. They will continue with the heart failure medications

INTERVENTIONS:
Procedure: Renal Denervation — Symplicity Catheter System
  Arms: Renal Denervation

SUMMARY:
The REACH study, is a prospective, double-blinded, randomised, controlled study of the safety and effectiveness of renal denervation in subjects with chronic systolic heart failure. Bilateral denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radio frequency (RF) energy through the luminal surface of the renal artery.

DETAILED DESCRIPTION:
Interventional study

Allocation: Randomised Endpoint Classification: Safety / Efficacy Study Intervention Model: Parallel Assignment Masking: Double blind (Subject / CHF team). The interventional operator, will have no role in care of the patient following randomisation.

Primary Purpose: Treatment

Chronic Systolic Heart Failure

Device: Renal denervation (Symplicity Catheter System) Symplicity Catheter System

-Intervention: Device: Renal denervation (Symplicity Catheter System)

Patients are randomised in the cath lab to receive either renal denervation or sham procedure.

Experimental arm: Renal Denervation Control arm: No renal denervation (sham procedure)

In both arms, aftercare is provided by clinicians who are blinded to the randomised allocation arm. Subjects will have been recruited on stable heart failure therapy, and the intention is to maintain this therapy steady during followup.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure due to systolic dysfunction
* New York Heart Association class II or higher
* Maximal pharmacological therapy including (where clinically indicated and tolerated), b-blocker, ACE inhibitors /A2 blocker, Aldosterone blockade.
* Ejection fraction less than 40%

Exclusion Criteria:

* Estimated GFR<35ml/hr
* Unfavourable renal anatomy (renal artery stenosis)
* Unable to walk on a treadmill for cardiopulmonary exercise test
* Significant valvular disease (moderate or more aortic regurgitation/stenosis or mitral stenosis; severe mitral/tricuspid regurgitation)
* Severe lung disease
* Symptomatic orthostatic dizziness
* Unable to consent
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in symptomatology | Baseline to 12 months post-randomization
  Improvement in symptomatology assessed using Kansas City Cardiomyopathy Questionnaire

SECONDARY OUTCOMES:
Improvement in peak VO2 on cardiopulmonary exercise testing | Baseline to 12 months post-randomization
  The peak VO2 will be compared in the interventional against the sham arm
Improvement in self-paced exercise distance | Baseline to 12 months post-randomization
  Improvement in 6 min walk to in interventional arm compared to sham arm
Change in chemoreflex sensitivity | Baseline to 12 months post-randomization
  Assess the change in chemoreflex sensitivity in the interventional arm in comparison to the sham arm
Change in NYHA functional classification | Baseline to 12 months post-randomization
  Assess the change in NYHA in interventional arm in comparison to sham arm
Incidence of Major Adverse Events | Baseline to 12 months post-randomization
  The incidence of major adverse events will be compared in the interventional against the sham arm

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, BA, MD, Study Director — Imperial College London; Justin E Davies, MBBS, PHD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Sobotka PA, Krum H, Bohm M, Francis DP, Schlaich MP. The role of renal denervation in the treatment of heart failure. Curr Cardiol Rep. 2012 Jun;14(3):285-92. doi: 10.1007/s11886-012-0258-x. PMID 22392370